CLINICAL TRIAL: NCT07214961
Title: Study to Investigate the Safety, Tolerability, Pharmacokinetics, Biodistribution and Antitumour Activity of the Alpha Radioligand Therapy AB001 in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Study of Alpha Radioligand Therapy AB001 in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Acronym: ARTISAN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ARTBIO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB001-101; 2024-516523-14 (EudraCT Number)
Record Dates: First submitted 2025-07-21; First posted 2025-10-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer (CRPC); Metastatic Castrate Resistant Prostate Cancer (mCRPC)
Keywords: radioligand therapy; Pb-212; castrate-resistant prostate cancer; alpha particles; metastatic; mCRPC; Lu-177
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: This is an open-label, noncontrolled, multinational, multicentre, interventional Phase 1 clinical study of AB001 in patients with advanced mCRPC.
  The study includes the following main parts:
  Dose Escalation: To assess the safety and tolerability of AB001 and determine the recommended dose level and treatment schedule in both 177Lu-PSMA naïve and 177Lu-PSMA experienced groups to take into the Expansion part.
  Dose Expansion: To further characterise the antitumour activity and safety profile of the recommended dose and schedule in both 177Lu-PSMA naïve and 177Lu-PSMA experienced groups for further development of AB001 in specific patient populations.
  Dose Escalation will seamlessly progress into Dose Expansion.
  The study will include several sub-studies to enable characterisation of the biodistribution, body clearance, and PK of AB001 in participants with mCRPC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AB001 treated ¹⁷⁷Lu-PSMA naïve mCRPC patients (Experimental): Dose Escalation will be initiated in ¹⁷⁷Lu-PSMA naïve mCRPC patients with the first cohort of participants receiving a starting dose of 100 MBq Pb212 (AB001) administered by slow injection on Day 1 of a 6-week (42-day) cycle. Four cycles of study treatment are planned; however, individual participants may continue up to a maximum of six treatment cycles provided they meet defined criteria. Subsequent cohorts of 177Lu-PSMA naïve participants will be opened for dose finding and schedule optimisation.
  Interventions: Drug: AB001
- AB001 treated 177Lu-PSMA experienced mCRPC patients (Experimental): For the 177Lu-PSMA experienced Group, the first cohort will initiate enrolment with a starting dose of 100 MBq Pb212 (AB001) administered by slow injection on Day 1 of a 6-week (42-day) cycle. Four cycles of study treatment are planned; however, individual participants may continue up to a maximum of six treatment cycles provided they meet defined criteria. Subsequent cohorts of 177Lu-PSMA experienced participants will be opened for dose finding and schedule optimisation.
  Interventions: Drug: AB001

INTERVENTIONS:
Drug: AB001 — Pb-212 PSMA targeted alpha radioligand therapy

SUMMARY:
This Phase 1 study will evaluate the safety, tolerability, and preliminary effectiveness of AB001, an alpha-emitting radioligand targeting prostate-specific membrane antigen (PSMA), in patients with advanced prostate cancer who are either 177Lu-PSMA naïve or experienced. The study includes dose escalation to identify a recommended dose and dose expansion to further assess safety and anti-tumour activity. Primary objectives are to characterize the safety profile and determine the optimal dose and schedule for future studies

ELIGIBILITY:
Inclusion Criteria:

* Male participants at least 18 years of age
* ECOG PS of 0 to 2
* Progressive mCRPC
* Previous treatment with at least one novel ARPI
* Prior orchiectomy and/or prior or ongoing androgen-deprivation therapy
* Prior treatment with at least one taxane regimen or patient refusing or considered appropriate by treating physician to delay taxane therapy
* 177Lu-PSMA experienced Group only: Prior treatment with at least one dose of 177Lu-PSMA
* At least one PSMA-avid distant metastatic lesion
* Adequate bone marrow, renal, and hepatic function

Exclusion Criteria

* Blockage in the bladder or kidneys
* Untreated or uncontrolled brain metastases. Treated brain metastases are permitted provided they are neurologically stable
* Symptomatic, or clinical or radiologic findings indicative of impending cord compression.
* History of myelodysplastic syndrome (MDS), treatment-related acute myeloid leukaemia or features suggestive of MDS/acute myeloid leukaemia.
* A known additional malignancy that has required active treatment within the past two years before start of study treatment, except for adequately treated basal or squamous cell carcinoma of the skin, or carcinoma in situ that has undergone curative therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-11-03 (Estimated); Study Completion 2028-11-03 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and tolerability profile of AB001 in participants with mCRPC | From enrolment to active follow-up at 12 months post end of treatment
  Incidence and severity of TEAEs (including AESIs and TESAEs)
Dose Escalation: To determine recommended AB001 Dose (MBq) in both 177Lu-PSMA naïve and 177Lu-PSMA experienced participants for Dose Expansion | For 177Lu-PSMA naïve group: Anticipated after 20 evaluable participants; ~1 year from FPFV in this group. For 177Lu-PSMA experienced group: Anticipated after 20 evaluable participants, ~1 year from FPFV in this group
  The recommended dose (MBq) of AB001 for dose expansion in 177Lu-PSMA naïve and experienced groups, determined based on safety and preliminary antitumour activity assessments (including incidence of DLTs and PSA50 response). The multiple measurements will be aggregated by the study team to select a single recommended dose.
  Single Outcome Measure Value (Units): Dose in MBq
Dose Escalation: To determine recommended AB001 Schedule (frequency of dose in cycles/weeks) in both 177Lu-PSMA naïve and 177Lu-PSMA experienced participants for Dose Expansion | Time Frame- For 177Lu-PSMA naïve group: Anticipated after 20 evaluable participants; ~1 year from FPFV in this group. For 177Lu-PSMA experienced group: Anticipated after 20 evaluable participants, ~1 year from FPFV in this group
  The recommended AB001 Schedule (frequency of dose in cycles/weeks) for dose expansion in 177Lu-PSMA naïve and experienced groups, determined based on safety and preliminary antitumour activity assessments (including incidence of DLTs and PSA50 response). The multiple measurements will be aggregated by the study team to select a single recommended AB001 Schedule.
  Single Outcome Measure Value (Units): AB001 Schedule in Cycles/weeks
Dose Expansion: To assess the recommended Dose (MBq) determined in Dose Escalation in both 177Lu-PSMA naïve and 177Lu-PSMA experienced participants for further clinical development of AB001 | In each group treated with selected dose, anticipated after 20 evaluable participants, ~1 year from FPFV in each group.
  The recommended dose (MBq) of AB001 for further clinical development of AB001 in 177Lu-PSMA naïve and experienced groups, determined based on safety and preliminary antitumour efficacy (including incidence and severity of [S]AEs, PSA50 response, and ORR). The multiple measurements will be aggregated by the study team to select a single recommended dose.
  Single Outcome Measure Value (Units): Dose in MBq
Dose Expansion: To assess the recommended AB001 Schedule (frequency of dose in cycles/weeks) determined in Dose Escalation in both 177Lu-PSMA naïve and 177Lu-PSMA experienced participants for further clinical development of AB001 | In each group treated with selected schedule, anticipated after 20 evaluable participants, ~1 year from FPFV in each group.
  The recommended schedule of AB001 for further clinical development of AB001 in 177Lu-PSMA naïve and experienced groups, determined based on safety and preliminary antitumour efficacy (including incidence and severity of [S]AEs, PSA50 response, and ORR). The multiple measurements will be aggregated by the study team to select a single recommended schedule of AB001.
  Single Outcome Measure Value (Units): AB001 Schedule in Cycles/weeks

CONTACTS AND LOCATIONS:
Overall Officials: CMO, Study Chair — ARTBIO Inc.
Locations (3):
- United States (3):
  - BAMF Health, Grand Rapids, Michigan
  - XCancer, Omaha, Nebraska
  - United Theranostics, Princeton, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided
Decision regarding sharing of de-identified IPD will be made at a later date